CLINICAL TRIAL: NCT03608072
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Rising Oral Doses of BI 690517 in Healthy Japanese Male Subjects (double-blind, Randomised, Placebo-controlled Within Dose Groups)
Brief Title: A Study in Healthy Japanese Men to Test How Different Doses of BI 690517 Are Taken Up in the Body and How Well They Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 1378-0004
Record Dates: First submitted 2018-07-20; First posted 2018-07-31 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose group 1 (Experimental)
  Interventions: Drug: BI 690517; Drug: Placebo
- Dose group 2 (Experimental)
  Interventions: Drug: BI 690517; Drug: Placebo
- Dose group 3 (Experimental)
  Interventions: Drug: BI 690517; Drug: Placebo

INTERVENTIONS:
Drug: BI 690517 — 3 sequential dose groups
  Other Names: Vicadrostat
Drug: Placebo — 3 sequential dose groups

SUMMARY:
The primary objective of the trial is to investigate the safety and tolerability of BI 690517 in healthy Japanese male subjects following oral administration of multiple rising doses over 14 days.

Secondary objective is the exploration of the pharmacokinetic(s) (PK) and pharmacodynamic(s) (PD) of BI 690517 in healthy Japanese male subjects after multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Japanese ethnicity, according to the following criteria:

  -- born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 20 to 50 years (incl.)
* Body mass index (BMI) of 18.5 to 25.0 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who agree to minimize the risk of female partners becoming pregnant by fulfilling any of the following criteria starting from at least 30 days before the first administration of trial medication and until 90 days after trial completion:

  * Use of adequate contraception, e.g. any of the following methods plus condom:

    --- combined oral contraceptives, intrauterine device
  * Vasectomised (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilised (including hysterectomy) of the subject's female partner

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy and/or surgery of the gastrointestinal tract that could interfere with the pharmacokinetics (PK) of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including human immunodeficiency virus (HIV), viral hepatitis, syphilis and/or tuberculosis or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold (or T-SPOT) test. (Subject with positive Hepatitis B core antibody will not allowed to participate in the study)
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QT interval corrected for heart rate using the method of Fridericia (QTcF) or Bazett (QTc interval prolongation))
* Participation in another trial where an investigational drug has been administered within 60 days or 5 half-lives (whichever is greater) prior to planned administration of trial medication, or current participation in another trial involving administration of investigational drug
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 200 mL within 30 days or 400 mL within 12 weeks prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within 1 week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Serum potassium levels >5.0 mmol/L (5.0 mEq/L) or serum sodium levels <135 mmol/L (135 mEq/L) in non-hemolysed blood at screening

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Number [N (%)] of subjects with drug-related adverse events (AEs) | Up to day 19

SECONDARY OUTCOMES:
AUCτ,1 (area under the concentration-time curve of the analyte in plasma over a uniform dosing interval τ after administration of the first dose [AUCτ,1 will be AUC0-24]) | up to 24 hours
Cmax (maximum measured concentration of the analyte in plasma) | Up to 24 hours
AUCτ,ss (area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ) | After 312 hours and up to 360 hours
Cmax,ss (maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ) | After 312 hours and up to 360 hours

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: Undecided
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions: 1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). Requestors can use the following link http:// trials.boehringer-ingelheim.com/ to:
  1. find information in order to request access to clinical study data, for listed studies.
  2. request access to clinical study documents that meet criteria, and upon a signed 'Document Sharing Agreement'.